CLINICAL TRIAL: NCT00444678
Title: A Phase II Study of Cetuximab Plus Biweekly Capecitabine and Oxaliplatin (C-CO2) in the Treatment of Patients With KRAS Wild Type Metastatic Colorectal Cancer
Brief Title: Cetuximab Plus Biweekly Capecitabine and Oxaliplatin in KRAS Wild Type Metastatic Colorectal Cancer
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: NYU Langone Health (Other)
Collaborators: Eli Lilly and Company (Industry); Bristol-Myers Squibb (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: NYU# 04-10 H11817; CA225056 (Other: Bristol-Myers Squibb)
Record Dates: First submitted 2007-03-07; First posted 2007-03-08 (Estimated); Results first posted 2020-04-03 (Actual); Last update posted 2020-04-03 (Actual); Status verified 2020-04

CONDITIONS: Colorectal Cancer; Neoplasm Metastasis
Keywords: Previously untreated metastatic colorectal cancer; Metastatic Colorectal Cancer; combined therapy; biologics therapy; antibody; chemotherapy; EGFR; epidermal growth factor receptor
MeSH Terms: conditions — Colorectal Neoplasms; Neoplasm Metastasis | interventions — Cetuximab; Oxaliplatin; Capecitabine

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No | US Export: No

ARMS (1):
- Cetuximab, Capecitabine and Oxaliplatin (Experimental)
  Interventions: Drug: Cetuximab; Drug: Oxaliplatin; Drug: Capecitabine

INTERVENTIONS:
Drug: Cetuximab — 500 mg/m2, IV every two weeks
  Other Names: Erbitux; C225
Drug: Oxaliplatin — 85 mg/m2, IV, q 2 weeks
  Other Names: Eloxatin
Drug: Capecitabine — 2500 mg, po bid x 7 days every two weeks
  Other Names: Xeloda

SUMMARY:
This is a Phase II, open label, non-randomized study in subjects with histologically confirmed diagnosis of advanced KRAS wild type adenocarcinoma of the colon or rectum, who have not received prior chemotherapy for metastatic disease.

DETAILED DESCRIPTION:
The current treatment options for metastatic colon cancer are in need of further improvement. The three-drug combination of oxaliplatin with 5-FU/LV (fluorouracil/leucovorin) in the second-line treatment of metastatic colorectal cancer have shown a significant increase in response rate compared to 5-FU/LV alone. Oxaliplatin has recently been FDA-approved for this indication and is now a standard first-line agent in combination with a fluoropyrimidine. Cetuximab, a chimeric monoclonal antibody against the growth factor receptor, has shown activity with and without irinotecan in subjects with colorectal cancer refractory to irinotecan alone. Cetuximab has also been shown to be safe and effective when administered with infusional 5-FU/folinic acid plus irinotecan. These results suggest that the addition of cetuximab to fluoropyrimidine/oxaliplatin-based regimen in the 1st line setting should be explored. The use of the oral fluoropyrimidine, capecitabine, to replace infusional 5FU has been widely used for improved convenience and possible safety. We have chosen a modified biweekly CapeOx (capecitabine plus oxaliplatin) regimen due to its improved tolerance and response rate with a fixed dose of capecitabine given its widespread practice and ease of use.

ELIGIBILITY:
Inclusion Criteria:

* Subjects must have signed an approved informed consent.
* Histologically confirmed diagnosis of advanced adenocarcinoma of the colon or rectum, with KRAS wild type on mutational analysis.
* No prior chemotherapy for metastatic disease (chemotherapy naive). Prior adjuvant therapy with 5FU/LV or IFL (irinotecan, fluorouracilis, and leucovorin (folinic acid)) permitted if completed at least six months prior to entering this study.
* Measurable disease by RECIST criteria as defined in Section 3.3.1.
* Subjects for whom tumor tissue is available for IHC ( Immunohistochemistry) testing for EGFR expression.
* ECOG (Eastern Cooperative Oncology Group) Performance Status 0-1.
* Recovery in full from any previous surgical procedure.
* Expected survival greater than 12 weeks.
* Subjects at least 18 years of age.
* Women of childbearing potential (WOCBP) must be using an adequate method of contraception to avoid pregnancy throughout the study and for up to 4 weeks after the study in such a manner that the risk of pregnancy is minimized. WOCBP must have a negative serum or urine pregnancy test (minimum sensitivity 25 IU/L or equivalent units of HCG) within 72 hours prior to the start of study medication.
* Adequate hematologic function defined by an absolute neutrophil count (ANC) > 1,500/mm3, a platelet count > 100,000/mm3 .
* Adequate hepatic function defined by a total bilirubin level no greater than 2.0 times the upper limit of normal (ULN) and AST (Aspartate Aminotransferase) and ALT (alanine transaminase) levels noo greater than 2.5 times the ULN (AST and ALT levels no greater than 5 times the ULN in the presence of liver metastases).
* Adequate renal function defined by a serum creatinine level no greater than 1.5 times the ULN.

Exclusion Criteria:

* WOCBP who are unwilling or unable to use an acceptable method to avoid pregnancy for the entire study period and for up to 4 weeks after the study.
* Women who are pregnant or breastfeeding.
* Women with a positive pregnancy test on enrollment or prior to study drug administration.
* Sexually active fertile men not using effective birth control if their partners are women of child-bearing potential.
* Subjects with > Grade 1 neuropathy.
* Any active or uncontrolled infection.
* History of myocardial infarction within the previous six months or current clinical evidence of congestive heart failure.
* History of any other cancer (except nonmelanoma skin cancer or carcinoma in situ of the cervix) unless in complete remission and off all therapy for that cancer for at least 5 years.
* Central nervous system metastases.
* Pregnant or lactating women. Men and women of reproductive potential must agree to use an effective contraceptive method.
* Medical or psychiatric disorders that would interfere with informed consent or make them a poor risk for participation in this trial.
* Prior allergic reaction to chimerized or murine monoclonal antibody therapy or documented presence of human anti-mouse antibodies (HAMA).
* Subjects receiving a prior investigational agent within 30 days.
* Prior therapy with oxaliplatin, cetuximab, or prior therapy that targets the EGF ( epidermal growth factor) pathway.
* Prisoners or subjects who are compulsorily detained (involuntarily incarcerated) for treatment of either a psychiatric or physical (e.g., infectious disease) illness must not be enrolled into this study.
* Mutation in the KRAS gene

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 36 (Actual)
Dates: Start 2004-06-01; Primary Completion 2012-08-01 (Actual); Study Completion 2015-06-01 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Deirdre Cohen, MD, Principal Investigator — NYU Langone Health
Locations (2):
- United States (2):
  - Bellevue Hospital, New York, New York
  - New York University Langone Medical Center, New York, New York

RESULTS

PARTICIPANT FLOW:
Period: Overall Study
Arm/Group | Cetuximab, Capecitabine and Oxaliplatin
Started | 36
Completed | 5
Not Completed | 31
Not completed — Toxicity | 11
Not completed — Disease Progression | 12
Not completed — Death | 3
Not completed — Physician Decision | 3
Not completed — Withdrawal by Subject | 2

BASELINE CHARACTERISTICS:
Arm/Group | Cetuximab, Capecitabine and Oxaliplatin
Number analyzed (Participants) | 36
Age, Continuous [Mean (Full Range); unit: years] | 62 [37 to 80]
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 15
  Male | 21
Race/Ethnicity, Customized [Count of Participants; unit: Participants]
  Asian | 7
  Black or African American | 3
  White | 21
  Unknown | 5
Region of Enrollment [Number; unit: participants]
  United States | 36

OUTCOME MEASURES:

1. Primary Outcome: Response Rate for the Combination Treatment
Description: The tumor response rate (RR) will be defined as the total number of subjects whose best response is partial response (PR) or complete response (CR) during the first six months of treatment, divided by the number of subjects.
Time Frame: 6 months since the start of treatment
Measure: Count of Participants; unit: Participants
Arm/Group | Cetuximab, Capecitabine and Oxaliplatin
Number analyzed (Participants) | 36
Participants | 21

2. Secondary Outcome: Toxicity Rates
Description: # of subjects who experienced >= grade 1 adverse event that is positively related to treatment.
Time Frame: 1 year since the first treatment and every year after for up to 10 years
Measure: Count of Participants; unit: Participants
Arm/Group | Cetuximab, Capecitabine and Oxaliplatin
Number analyzed (Participants) | 36
Participants | 36

3. Secondary Outcome: Time to Progression
Description: Time to Treatment Failure (progression or death) will be defined as the time from the first day of treatment until the date Progressive Disease (PD) or death is first reported. Subjects who die without a reported prior progression will be considered to have progressed on the day of their death. Subjects who did not progress will be censored at the day of their last tumor assessment.
Time Frame: 6 months since the start of treatment and every 3 months after treatment for up to 10 years
Measure: Median (Full Range); unit: Days
Arm/Group | Cetuximab, Capecitabine and Oxaliplatin
Number analyzed (Participants) | 36
Days | 275 [43 to 2822]

4. Secondary Outcome: Survival
Description: Survival will be defined as the number of days from the first day of therapy to the date of death. If the subject is lost to follow-up, survival will be censored on the last date the subject was known to be alive.
Time Frame: 6 months since the start of treatment and every 3 months after treatment for up to 10 years
Measure: Median (Full Range); unit: Days
Arm/Group | Cetuximab, Capecitabine and Oxaliplatin
Number analyzed (Participants) | 36
Days | 417 [43 to 4166]

ADVERSE EVENTS:
Time Frame: 3 years
Arm/Group | Cetuximab, Capecitabine and Oxaliplatin
All-Cause Mortality (participants affected / at risk) | 3/36
Serious Adverse Events (participants affected / at risk) | 14/36
Other Adverse Events (participants affected / at risk) | 26/36
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Cetuximab, Capecitabine and Oxaliplatin (N=36)
Shortness Of Breath (Respiratory, thoracic and mediastinal disorders) | 1 (1)
diarrhea (Gastrointestinal disorders) | 4 (4)
Vasovagal Episode (Cardiac disorders) | 1 (1)
hypotension (Cardiac disorders) | 1 (1)
dehydration (Gastrointestinal disorders) | 3 (3)
Nausea (Gastrointestinal disorders) | 2 (2)
seizure (Nervous system disorders) | 1 (1)
Vomiting (Gastrointestinal disorders) | 2 (2)
Thrombosis (Cardiac disorders) | 1 (1)
Death (Cardiac disorders) | 1 (1) — (Arrhythmia)
Obstruction - Gi (Gastrointestinal disorders) | 3 (3)
Hemorrage/ Bleeding (Blood and lymphatic system disorders) | 1 (1)
fatigue (General disorders) | 3 (3)
colitis (Gastrointestinal disorders) | 1 (1)
Infection (Immune system disorders) | 2 (2)
Cardiopulmonary Arrest (Cardiac disorders) | 1 (1)
Sepsis (Infections and infestations) | 2 (2)
Fistula (Gastrointestinal disorders) | 1 (1)
Abdominal Pain (Gastrointestinal disorders) | 2 (2)
Anorexia (Gastrointestinal disorders) | 1 (1)
Weight loss (Metabolism and nutrition disorders) | 1 (1)
Disease progression on study (Gastrointestinal disorders) | 1 (1)
OTHER ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | Cetuximab, Capecitabine and Oxaliplatin (N=36)
Abdominal pain or cramping (Gastrointestinal disorders) | 12
Alkaline phosphatase (General disorders) | 3
Allergic reaction/hypersensitivity (including drug fever) (General disorders) | 1
Alopecia (Skin and subcutaneous tissue disorders) | 1
Anorexia (Psychiatric disorders) | 18
Arthralgia (joint pain) (Musculoskeletal and connective tissue disorders) | 1
Ascites (non-malignant) (Gastrointestinal disorders) | 1
Bicarbonate (Renal and urinary disorders) | 2
bilirubin (Hepatobiliary disorders) | 1
Blood/Bone Marrow-Other (Blood and lymphatic system disorders) | 1
Bruising (in absence of grade 3 or 4 thrombocytopenia) (Blood and lymphatic system disorders) | 1
Cardiovascular/Arrhythmia-Other (Cardiac disorders) | 2
Colitis (Gastrointestinal disorders) | 2
Constipation (Gastrointestinal disorders) | 11
Constitutional Symptoms-Other (General disorders) | 2
Cough (Respiratory, thoracic and mediastinal disorders) | 2
Dehydration (General disorders) | 4
Dermatology/Skin-Other (Skin and subcutaneous tissue disorders) | 12
Diarrhea - patients with a colostomy (Gastrointestinal disorders) | 3
Diarrhea - patients without colostomy (Gastrointestinal disorders) | 20
Dizziness/lightheadedness (Nervous system disorders) | 5
Dry Eye (Eye disorders) | 1
Dry Skin (Skin and subcutaneous tissue disorders) | 4
Dyspepsia/heartburn (Gastrointestinal disorders) | 5
Dysphagia, esophagitis, odynophagia (painful swallowing) (General disorders) | 2
Dyspnea (shortness of breath) (Respiratory, thoracic and mediastinal disorders) | 5
Dysuria (painful urination) (Renal and urinary disorders) | 1
Edema (Blood and lymphatic system disorders) | 3
Erectile impotence (Reproductive system and breast disorders) | 1
Fatigue (lethargy, malaise, asthenia) (General disorders) | 20
Febrile neutropenia (Immune system disorders) | 1
Fever (in the absence of neutropenia) (General disorders) | 5
Fistula-intestinal (Gastrointestinal disorders) | 1
Flatulence (Gastrointestinal disorders) | 5
Flushing (General disorders) | 1
Gastrointestinal-Other (Gastrointestinal disorders) | 6
Nausea (General disorders) | 26
Rash/desquamation (Skin and subcutaneous tissue disorders) | 25
Neuropathy-sensory (Nervous system disorders) | 22
Stomatitis/pharyngitis (oral/pharyngeal mucositis) (General disorders) | 17

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: Yes